CLINICAL TRIAL: NCT03046056
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled Study Evaluating the Efficacy and Safety of Filgotinib in the Treatment of Small Bowel Crohn's Disease (SBCD)
Brief Title: Study to Evaluate the Efficacy and Safety of Filgotinib in the Treatment of Small Bowel Crohn's Disease (SBCD)
Acronym: DIVERGENCE 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-419-4015; 2016-003179-23 (EudraCT Number)
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Results first posted 2021-08-09 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Small Bowel Crohn's Disease
MeSH Terms: interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Filgotinib 200 mg (Experimental): Filgotinib 200 mg tablet + placebo to match (PTM) filgotinib 100 mg tablet for up to 27 weeks.
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib
- Filgotinib 100 mg (Experimental): Filgotinib 100 mg tablet + PTM filgotinib 200 mg tablet for up to 26.3 weeks.
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib
- Placebo (Placebo Comparator): PTM filgotinib 200 mg tablet + PTM filgotinib 100 mg tablet for up to 28.7 weeks.
  Interventions: Drug: Placebo to match filgotinib

INTERVENTIONS:
Drug: Filgotinib — Tablet(s) administered orally once daily
  Other Names: GS-6034; GLPG0634
  Arms: Filgotinib 100 mg; Filgotinib 200 mg
Drug: Placebo to match filgotinib — Tablet(s) administered orally once daily

SUMMARY:
The primary objective of this study is to evaluate the efficacy of filgotinib, when compared to placebo, in establishing clinical remission defined as Crohn's disease activity index (CDAI) < 150, at Week 24 in participants with small bowel Crohn's disease (CD). Participants will have the option to enter a separate long-term extension study if they meet eligibility requirements.

ELIGIBILITY:
Key Inclusion Criteria:

* Males or non-pregnant, nonlactating females, ages 18 to 75 years, inclusive based on the date of screening visit
* Moderately or severely active CD
* Minimum duration of CD of at least 6 months
* Presence of diseased small bowel (SB) segments in at least 1 of the following segments: terminal ileum, distal ileum, or jejunum
* Patients with additional colonic involvement of CD are permitted in study as long as SBCD is present
* Previously demonstrated an inadequate clinical response, loss of response to, or intolerance to at least 1 of the following agents (depending on current country treatment recommendations/guidelines):

  * Corticosteroids
  * Immunomodulators
  * Tumor necrosis factor-alpha (TNFα) antagonists
  * Vedolizumab
  * Ustekinumab
* Willing and able to undergo magnetic resonance enterography (MRE) per protocol requirements

Key Exclusion Criteria:

* Presence of symptomatic or clinically significant (eg, obstructive or symptomatic) strictures or stenosis.
* Presence of fistulae
* Evidence of short bowel syndrome
* Presence of ulcerative colitis, indeterminate colitis, ischemic colitis, fulminant colitis, or toxic mega-colon
* History of total colectomy, subtotal-colectomy, presence of ileostomy or colostomy, or likely requirement for surgery during the study
* Use of any prohibited concomitant medications as described in the study protocol
* Active tuberculosis (TB) or history of latent TB that has not been treated

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (38):
- United States (15):
  - University of Miami Crohn's and Colitis Center, Miami, Florida
  - Center for lnterventional Endoscopy- Florida Hospital, Orlando, Florida
  - University of South Florida South Tampa campus, Tampa, Florida
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Gastro Center of Maryland, Columbia, Maryland
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - Fargo Gastroenterology and Hepatology Clinic, Fargo, North Dakota
  - Gastro One, Germantown, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - TDDC San Marcos, San Marcos, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - McGuire DVAMC, Richmond, Virginia
- Austria (2):
  - Medical University of Innsbruck, Department of Internal Medicine I, Innsbruck
  - Medical University of Vienna, Department of Internal Medicine III, Division Gastroenterology and Hepatology, Vienna
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Centre Hospitalier Chretien, Liège
- Canada (2):
  - Mount Sinai Hospital, Toronto
  - PerCuro Clinical Research Ltd., Victoria
- Hepato-Gastroenterologie HK, s.r.o., Hradec Králové, Czechia
- CHU de Toulouse -Hopital Rangueil (Main Office), Toulouse, Midi-Pyrenees, France
- Germany (2):
  - Gastroenterologie, Hepatologie und Endokrinologie, Hanover
  - Universitatsklinikum Jena, Jena
- Hungary (2):
  - Bugát Pál Kórház, Gasztroenterológiai osztály, Gyöngyös, Heves County
  - Békés Megyei Központi Kórház Dr. Réthy Pál Tagkórháza, Békéscsaba
- Italy (2):
  - Azienda Ospedaliero - Universitaria Mater Domini, Catanzaro
  - Gastroenterologia, Policlinico Universitario Campus Bio-Medico di Roma, Rome
- Spain (2):
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
- Ukraine (3):
  - Ivano-Frankivsk Central City Clinical Hospital, Department of Therapy #1, SHEI Ivano-Frankivsk National Medical University, Ivano-Frankivsk
  - Communal Healthcare Institution Regional Hospital of War Veterans, Department of Therapy #1, Kharkiv
  - Communal Institution of Ternopil Regional Council Ternopil University Hospital. Regional Center of Gastroenterology, Ternopil
- United Kingdom (4):
  - Queen Elizabeth University Hospital, Glasgow, Scotland
  - Royal Devon and Exeter Hospital, Department of Gastroenterology, Exeter
  - St Georges Clinical Research Facility, London
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riviere P, D'Haens G, Peyrin-Biroulet L, Baert F, Lambrecht G, Pariente B, Bossuyt P, Buisson A, Oldenburg B, Vermeire S, Laharie D. Location but Not Severity of Endoscopic Lesions Influences Endoscopic Remission Rates in Crohn's Disease: A Post Hoc Analysis of TAILORIX. Am J Gastroenterol. 2021 Jan 1;116(1):134-141. doi: 10.14309/ajg.0000000000000834. PMID 33177349

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Canada, and Europe. The first participant was screened on 11 April 2017. The last study visit occurred on 20 July 2020.
Pre-assignment Details: 198 participants were screened.
Groups:
- Filgotinib 200 mg: Filgotinib 200 mg tablet + placebo to match (PTM) filgotinib 100 mg tablet orally once daily for up to 27 weeks.
- Filgotinib 100 mg: Filgotinib 100 mg tablet + PTM filgotinib 200 mg tablet orally once daily for up to 26.3 weeks.
- Placebo: PTM filgotinib 200 mg tablet + PTM filgotinib 100 mg tablet orally once daily for up to 28.7 weeks.
Period: Overall Study
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Started | 28 | 32 | 18
Completed | 16 | 16 | 11
Not Completed | 12 | 16 | 7
Not completed — Non-responder at Week 10 | 6 | 6 | 4
Not completed — Protocol-specified Disease Worsening | 3 | 3 | 1
Not completed — Adverse Event | 1 | 5 | 0
Not completed — Non-compliance With Study Drug | 0 | 0 | 2
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Investigator's Discretion | 0 | 1 | 0
Not completed — Withdrew Consent | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Filgotinib 200 mg: Filgotinib 200 mg tablet + PTM filgotinib 100 mg tablet orally once daily for up to 27 weeks.
- Total: Total of all reporting groups
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo | Total
Number analyzed (Participants) | 28 | 32 | 18 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (16.3) | 42 (12.9) | 45 (12.9) | 44 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 9 | 51
  Male | 9 | 9 | 9 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted means local regulators did not allow collection of race information.
  Participants
    Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Race: Asian | 0 | 0 | 0 | 0
    Race: Black or African American | 2 | 4 | 2 | 8
    Race: Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0
    Race: White | 25 | 28 | 16 | 69
    Race: Other | 1 | 0 | 0 | 1
    Race: Not Permitted | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted means local regulators did not allow collection of ethnicity information.
  Participants
    Ethnicity: Not Hispanic or Latino | 26 | 31 | 17 | 74
    Ethnicity: Hispanic or Latino | 2 | 1 | 1 | 4
    Ethnicity: Not Permitted | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 13 | 10 | 38
  Hungary | 0 | 3 | 1 | 4
  Czechia | 0 | 1 | 0 | 1
  Ukraine | 2 | 0 | 1 | 3
  United Kingdom | 4 | 1 | 2 | 7
  Spain | 1 | 2 | 0 | 3
  Canada | 0 | 4 | 1 | 5
  Austria | 1 | 1 | 0 | 2
  Belgium | 0 | 2 | 0 | 2
  Italy | 3 | 1 | 1 | 5
  France | 2 | 2 | 1 | 5
  Germany | 0 | 2 | 1 | 3
Crohn's Disease Activity Index Score (CDAI) [Mean (Standard Deviation); unit: score on scale] — The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. The score ranges from 0 to 600. A score of < 150 indicates remission. A higher score indicates more severe disease.
  score on scale | 309 (55.7) | 297 (64.9) | 300 (63.7) | 302 (60.9)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Clinical Remission at Week 24
Description: The CDAI score is used to quantify the symptoms of participants with Crohn's Disease (CD). The score ranges from 0 to 600. Clinical remission by CDAI was defined as a score of < 150. A higher score indicates more severe disease.
Time Frame: Week 24
Population: Full Analysis Set included all the randomized participants who received at least one dose of the study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 28 | 32 | 18
percentage of participants | 25.0 [12.4 to 41.9] | 25.0 [13.1 to 40.6] | 16.7 [4.7 to 37.7]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Test type: Superiority; Risk Difference in Proportions = 8.3, 90% CI 2-sided [-16.5 to 32.1]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Test type: Superiority; Risk Difference in Proportions = 8.3, 90% CI 2-sided [-15.9 to 32.0]

2. Secondary Outcome: Change From Baseline in Terminal Ileum Segmental Magnetic Resonance Index of Activity (MaRIA) Score at Week 24
Description: Magnetic resonance enterography (MRE) is an imaging technique to evaluate disease activity in CD. MaRIA is an MRE-based scoring system. The MaRIA scoring system is a composite index of 4 components. These components are edema, ulcers, gut wall thickness, and relative contrast enhancement (RCE). A segmental MaRIA score can be calculated at screening (used as the baseline) and Week 24 as a weighted sum of these components for the terminal ileum segment of the small bowel. A segmental score of ≥ 7 indicates active inflammation and a score of ≥ 11 indicates the presence of an ulcer. Segmental scores less than 7 indicate remission. The MaRIA score ranges from approximately 0 to 31, for any given segment. A higher score indicates more severe disease. Difference in least squared means (Diff in LSM) were from analysis of covariance (ANCOVA) model. A negative change from baseline indicates improvement and a positive change from baseline indicates disease worsening.
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 28 | 32 | 18
score on scale | -1.8 (1.51) | 0.7 (1.39) | 0.5 (1.64)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Difference in least squared means (Diff in LSM), and its 90% confidence interval (CI) were from analysis of covariance (ANCOVA) model adjusted by baseline segmental MaRIA score, concomitant use of oral, systemically absorbed corticosteroids at baseline, concomitant use of immunomodulators at baseline, prior exposure to biologics, and treatment group; Test type: Superiority; Least Squares Mean Difference = -2.3, 90% CI 2-sided [-5.3 to 0.7], Standard Error of Mean 1.81
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Diff in LSM, and its 90% CI were from ANCOVA model adjusted by baseline segmental MaRIA score, concomitant use of oral, systemically absorbed corticosteroids at baseline, concomitant use of immunomodulators at baseline, prior exposure to biologics, and treatment group; Test type: Superiority; Least Squares Mean Difference = 0.2, 90% CI 2-sided [-2.7 to 3.1], Standard Error of Mean 1.72

3. Secondary Outcome: Change From Baseline in Distal Ileum Segmental MaRIA Score at Week 24
Description: MRE is an imaging technique to evaluate disease activity in CD. MaRIA is an MRE-based scoring system. The MaRIA scoring system is a composite index of 4 components. These components are edema, ulcers, gut wall thickness, and RCE. A segmental MaRIA score can be calculated at Screening (used as the baseline) and Week 24 as a weighted sum of these 4 components for the distal ileum segment of the small bowel. A segmental score of ≥ 7 indicates active inflammation and a score of ≥ 11 indicates the presence of an ulcer. Segmental scores less than 7 indicate remission in that segment. The MaRIA score ranges from approximately 0 to 31, for any given segment. A higher score indicates more severe disease. Diff in LSM were from ANCOVA model. A negative change from baseline indicates improvement and a positive change from baseline indicates disease worsening.
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 28 | 32 | 18
score on scale | -1.1 (1.12) | -0.5 (1.08) | 0.5 (1.26)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Least Squares Mean Difference = -1.6, 90% CI 2-sided [-3.9 to 0.7], Standard Error of Mean 1.38
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Least Squares Mean Difference = -1.0, 90% CI 2-sided [-3.2 to 1.2], Standard Error of Mean 1.32

4. Secondary Outcome: Change From Baseline in Jejunum Segmental MaRIA Score at Week 24
Description: MRE is an imaging technique to evaluate disease activity in CD. MaRIA is an MRE-based scoring system.The MaRIA scoring system is a composite index of 4 components. These components are edema, ulcers, gut wall thickness, and RCE. A segmental MaRIA score can be calculated at Screening (used as the baseline) and Week 24 as a weighted sum of these 4 components for the jejunum segment of the small bowel. A segmental score of ≥ 7 indicates active inflammation and a score of ≥ 11 indicates the presence of an ulcer. Segmental scores less than 7 indicate remission in that segment. The MaRIA score ranges from approximately 0 to 31, for any given segment. A higher score indicates more severe disease. Diff in LSM were from ANCOVA model. A positive change from baseline indicates disease worsening.
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 28 | 32 | 18
score on scale | 0.4 (1.00) | 0.6 (0.95) | 0.5 (1.12)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Least Squares Mean Difference = -0.1, 90% CI 2-sided [-2.2 to 2.0], Standard Error of Mean 1.24
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Least Squares Mean Difference = 0.1, 90% CI 2-sided [-1.9 to 2.0], Standard Error of Mean 1.18

5. Secondary Outcome: Percentage of Participants Who Achieved MaRIA Remission in Terminal Ileum Segment at Week 24
Description: The MaRIA scoring system is a composite index of 4 components. These components are edema, ulcers, gut wall thickness, and RCE. A segmental MaRIA score can be calculated at screening (used as the baseline) and Week 24 as a weighted sum of these 4 components for the terminal ileum segment of the small bowel. The MaRIA score ranges from approximately 0 to 31, for any given segment. A higher score indicates more severe disease. MaRIA remission was defined as a segmental MaRIA score < 7 in terminal ileum segment at Week 24 among participants with MaRIA score ≥ 7 in the same segment at baseline. A segmental score of ≥ 7 indicates active inflammation and a score of ≥ 11 indicates the presence of an ulcer.
Time Frame: Week 24
Population: Participants in the Full Analysis Set with active disease (segmental MaRIA score ≥ 7) in terminal ileum segment at baseline, were analyzed.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 22 | 30 | 16
percentage of participants | 4.5 [0.2 to 19.8] | 6.7 [1.2 to 19.5] | 6.3 [0.3 to 26.4]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Test type: Superiority; Risk Difference in Proportions = -1.7, 90% CI 2-sided [-28.6 to 25.5]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Test type: Superiority; Risk Difference in Proportions = 0.4, 90% CI 2-sided [-24.5 to 26.2]

6. Secondary Outcome: Percentage of Participants Who Achieved MaRIA Remission in Distal Ileum Segment at Week 24
Description: The MaRIA scoring system is a composite index of 4 components. These components are edema, ulcers, gut wall thickness, and RCE. A segmental MaRIA score can be calculated at screening (used as the baseline) and Week 24 as a weighted sum of these 4 components for the distal ileum segment of the small bowel. The MaRIA score ranges from approximately 0 to 31, for any given segment. A higher score indicates more severe disease. MaRIA remission was defined as a segmental MaRIA score < 7 in distal ileum segment at Week 24 among participants with MaRIA score ≥ 7 in the same segment at baseline. A segmental score of ≥ 7 indicates active inflammation and a score of ≥ 11 indicates the presence of an ulcer.
Time Frame: Week 24
Population: Participants in the Full Analysis Set with active disease (segmental MaRIA score ≥ 7) in distal ileum segment at baseline, were analyzed.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 10 | 8 | 6
percentage of participants | 10.0 [0.5 to 39.4] | 0 [0.0 to 31.2] | 16.7 [0.9 to 58.2]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Test type: Superiority; Risk Difference in Proportions = -6.7, 90% CI 2-sided [-47.3 to 37.0]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Test type: Superiority; Risk Difference in Proportions = -16.7, 90% CI 2-sided [-58.2 to 30.0]

7. Secondary Outcome: Percentage of Participants Who Achieved MaRIA Remission in Jejunum Segment at Week 24
Description: The MaRIA scoring system is a composite index of 4 components. These components are edema, ulcers, gut wall thickness, and RCE. A segmental MaRIA score can be calculated at screening (used as the baseline) and Week 24 as a weighted sum of these 4 components for the jejunum segment of the small bowel. The MaRIA score ranges from approximately 0 to 31, for any given segment. A higher score indicates more severe disease. MaRIA remission was defined as a segmental MaRIA score < 7 in jejunum segment at Week 24 among participants with MaRIA score ≥ 7 in the same segment at baseline. A segmental score of ≥ 7 indicates active inflammation and a score of ≥ 11 indicates the presence of an ulcer.
Time Frame: Week 24
Population: Participants in the Full Analysis Set with active disease (segmental MaRIA score ≥ 7) in jejunum segment at baseline, were analyzed.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 6 | 8 | 3
percentage of participants | 33.3 [6.3 to 72.9] | 0 [0.0 to 31.2] | 0 [0.0 to 63.2]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Test type: Superiority; Risk Difference in Proportions = 33.3, 90% CI 2-sided [-32.4 to 86.5]

8. Secondary Outcome: Percentage of Participants Who Achieved MaRIA Response in Terminal Ileum Segment at Week 24
Description: The MaRIA scoring system is a composite index of 4 components. These components are edema, ulcers, gut wall thickness, and RCE. A segmental MaRIA score can be calculated at screening (used as the baseline) and Week 24 as a weighted sum of these 4 components for the terminal ileum segment of the small bowel. The MaRIA score ranges from approximately 0 to 31, for any given segment. A higher score indicates more severe disease. MaRIA response was defined as a segmental MaRIA score < 11 with baseline score ≥ 11, or a segmental MaRIA score < 7 with baseline score < 11, or ≥ minimum detectable difference (MDD) units decrease from baseline score for segments with baseline MaRIA score ≥ 7 in the terminal ileum. For segments with baseline MaRIA score ≥ 15, the MDD is 6.5 units and for baseline MaRIA score < 15, the MDD is 4.0 units.
Time Frame: Week 24
Population: as for outcome 5
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 22 | 30 | 16
percentage of participants | 22.7 [9.4 to 42.0] | 10.0 [2.8 to 23.9] | 25.0 [9.0 to 48.4]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Test type: Superiority; Risk Difference in Proportions = -2.3, 90% CI 2-sided [-28.6 to 24.3]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Test type: Superiority; Risk Difference in Proportions = -15.0, 90% CI 2-sided [-39.4 to 11.3]

9. Secondary Outcome: Percentage of Participants Who Achieved MaRIA Response in Distal Ileum Segment at Week 24
Description: The MaRIA scoring system is a composite index of 4 components. These components are edema, ulcers, gut wall thickness, and RCE. A segmental MaRIA score can be calculated at screening (used as the baseline) and Week 24 as a weighted sum of these 4 components for the distal ileum segment of the small bowel. The MaRIA score ranges from approximately 0 to 31, for any given segment. A higher score indicates more severe disease. MaRIA response was defined as a segmental MaRIA score < 11 with baseline score ≥ 11, or a segmental MaRIA score < 7 with baseline score < 11, or ≥ MDD units decrease from baseline score for segments with baseline MaRIA score≥ 7 in the distal ileum. For segments with baseline MaRIA score ≥ 15, the minimum detectable difference (MDD) is 6.5 units and for baseline MaRIA score < 15, the MDD is 4.0 units.
Time Frame: Week 24
Population: as for outcome 6
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 10 | 8 | 6
percentage of participants | 20.0 [3.7 to 50.7] | 12.5 [0.6 to 47.1] | 16.7 [0.9 to 58.2]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Test type: Superiority; Risk Difference in Proportions = 3.3, 90% CI 2-sided [-38.9 to 45.7]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Test type: Superiority; Risk Difference in Proportions = -4.2, 90% CI 2-sided [-47.5 to 40.8]

10. Secondary Outcome: Percentage of Participants Who Achieved MaRIA Response in Jejunum Segment at Week 24
Description: The MaRIA scoring system is a composite index of 4 components. These components are edema, ulcers, gut wall thickness, and RCE. A segmental MaRIA score can be calculated at screening (used as the baseline) and Week 24 as a weighted sum of these 4 components for the jejunum segment of the small bowel. The MaRIA score ranges from approximately 0 to 31, for any given segment. A higher score indicates more severe disease. MaRIA response was defined as a segmental MaRIA score < 11 with baseline score ≥ 11, or a segmental MaRIA score < 7 with baseline score < 11, or ≥ MDD units decrease from baseline score for segments with baseline MaRIA score ≥ 7 in the jejunum. For segments with baseline MaRIA score ≥ 15, the MDD is 6.5 units and for baseline MaRIA score < 15, the MDD is 4.0 units.
Time Frame: Week 24
Population: as for outcome 7
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 6 | 8 | 3
percentage of participants | 50.0 [15.3 to 84.7] | 12.5 [0.6 to 47.1] | 0 [0.0 to 63.2]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Test type: Superiority; Risk Difference in Proportions = 50.0, 90% CI 2-sided [-16.8 to 89.5]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Test type: Superiority; Risk Difference in Proportions = 12.5, 90% CI 2-sided [-46.1 to 63.3]

11. Secondary Outcome: Percentage of Participants Who Achieved Participant Level Small Bowel MaRIA Remission at Week 24
Description: The MaRIA scoring system is a composite index of 4 components. These components are edema, ulcers, gut wall thickness, and RCE. A segmental MaRIA score can be calculated at screening (used as the baseline) and Week 24 as a weighted sum of these 4 components for each of the 3 small bowel segments. The MaRIA score ranges from approximately 0 to 31, for any given segment. A higher score indicates more severe disease. Small bowel MaRIA remission was defined as MaRIA score < 7 at Week 24 in each of the 3 small bowel segments, among participants with MaRIA score ≥ 7 in at least 1 small bowel segment at baseline.
Time Frame: Week 24
Population: Participants in the Full Analysis Set with active disease (segmental MaRIA score ≥ 7) in at least 1 small bowel segment at baseline, were analyzed.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 25 | 32 | 18
percentage of participants | 8.0 [1.4 to 23.1] | 6.3 [1.1 to 18.4] | 0 [0.0 to 15.3]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Test type: Superiority; Risk Difference in Proportions = 8.0, 90% CI 2-sided [-17.2 to 32.6]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Test type: Superiority; Risk Difference in Proportions = 6.3, 90% CI 2-sided [-18.1 to 30.2]

12. Secondary Outcome: Percentage of Participants Who Achieved Participant Level Small Bowel MaRIA Response at Week 24
Description: The MaRIA scoring system is a composite index of 4 components. These components are edema, ulcers, gut wall thickness, and RCE. A segmental MaRIA score can be calculated at screening (used as the baseline) and Week 24 as a weighted sum of these 4 components for each of the 3 small bowel segments. The MaRIA score ranges from approximately 0 to 31, for any given segment. A higher score indicates more severe disease. Participant level small bowel MaRIA response was defined as all small bowel segments with baseline MaRIA score ≥7 achieve segment level MaRIA response, with no segment level disease worsening in any other segment(s) at Week 24, among participants with MaRIA score ≥ 7 in at least 1 small bowel segment at baseline.
Time Frame: Week 24
Population: as for outcome 11
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 25 | 32 | 18
percentage of participants | 20.0 [8.2 to 37.5] | 12.5 [4.4 to 26.4] | 16.7 [4.7 to 37.7]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Test type: Superiority; Risk Difference in Proportions = 3.3, 90% CI 2-sided [-22.1 to 28.1]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Test type: Superiority; Risk Difference in Proportions = -4.2, 90% CI 2-sided [-28.1 to 20.3]

13. Secondary Outcome: Percentage of Participants Who Achieved Early Clinical Remission by Crohn's Disease Activity Index (CDAI) at Week 10
Description: The CDAI score is used to quantify the symptoms of participants with CD. The score ranges from 0 to 600. Clinical remission by CDAI was defined as a score of < 150. A higher score indicates more severe disease.
Time Frame: Week 10
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 28 | 32 | 18
percentage of participants | 39.3 [23.8 to 56.5] | 25.0 [13.1 to 40.6] | 22.2 [8.0 to 43.9]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Test type: Superiority; Risk Difference in Proportions = 17.1, 90% CI 2-sided [-7.6 to 40.4]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Test type: Superiority; Risk Difference in Proportions = 2.8, 90% CI 2-sided [-21.2 to 26.5]

14. Secondary Outcome: Change From Baseline in CDAI Scores at Week 10
Description: The CDAI score is used to quantify the symptoms of participants with CD. The score ranges from 0 to 600. A score of < 150 indicates remission. A higher score indicates more severe disease. Difference in least squared means (Diff in LSM) were from analysis of covariance (ANCOVA) model. A negative change from baseline indicates improvement.
Time Frame: Baseline; Week 10
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 28 | 32 | 18
score on scale | -105 (23.6) | -88 (22.3) | -57 (26.2)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Least Squares Mean Difference = -48, 90% CI 2-sided [-95 to -1], Standard Error of Mean 28.1
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Least Squares Mean Difference = -31, 90% CI 2-sided [-76 to 15], Standard Error of Mean 27.4

15. Secondary Outcome: Change From Baseline in CDAI Scores at Week 24
Description: The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. The score ranges from 0 to 600. A score of < 150 indicates remission. A higher score indicates more severe disease. Diff in LSM were from ANCOVA model. A negative change from baseline indicates improvement.
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 28 | 32 | 18
score on scale | -86 (24.1) | -71 (22.8) | -66 (26.7)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Least Squares Mean Difference = -20, 90% CI 2-sided [-68 to 28], Standard Error of Mean 28.7
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Least Squares Mean Difference = -5, 90% CI 2-sided [-52 to 42], Standard Error of Mean 28.0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: First dose date up to last dose date (maximum: 28.7 weeks) plus 59 days; Adverse Events: First dose date up to last dose date (maximum: 28.7 weeks) plus 30 days
Description: All-Cause Mortality: All Randomized Analysis Set included all participants who were randomized in the study; Adverse Events: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/28 | 0/32 | 0/18
Serious Adverse Events (participants affected / at risk) | 4/28 | 7/32 | 0/18
Other Adverse Events (participants affected / at risk) | 20/28 | 24/32 | 13/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Filgotinib 200 mg (N=28) | Filgotinib 100 mg (N=32) | Placebo (N=18)
Crohn's disease (Gastrointestinal disorders) | 2 | 4 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Filgotinib 200 mg (N=28) | Filgotinib 100 mg (N=32) | Placebo (N=18)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 6 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 4 | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 5 | 3 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2
Asthenia (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 2 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 3 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 4 | 0
Sinusitis (Infections and infestations) | 4 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 2
Headache (Nervous system disorders) | 4 | 4 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 3 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT03046056/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT03046056/SAP_001.pdf